CLINICAL TRIAL: NCT03183583
Title: Tissue Adhesive in Hip and Knee Arthroplasty, A Cost -Effectiveness Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Amphia Hospital (Other)
Collaborators: R.C.I. van Geenen, orthopedic surgeon, Amphia, Breda, The Netherlands (Unknown); Ethicon, Inc. (Industry)
Responsible Party: Principal Investigator, Koen Koenraadt, coordinator FORCE, Amphia Hospital
Other Study IDs: IIS 15-212
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis
Keywords: Tissue Adhesive
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee | interventions — Tissue Adhesives; Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Tissue adhesive in primary Total Hip and Total Knee arthroplasty — Use of tissue adhesive in primary Total Hip and Total Knee arthroplasty

SUMMARY:
Prolonged wound drainage after total hip or knee arthroplasty is a very undesirable complication, both from medical as patients view. Wound drainage prolongs hospital admission and is associated with an increased risk of infection (1) post-operative wound drainage of more than 48 hours is associated with an increased infection risk of 42 percent a day in hip arthroplasty and 27 percent a day in knee arthroplasty. (2) Patient organizations report that wound drainage is considered as one of the most undesirable complications.

In our hospital, patients undergoing hip or knee arthroplasty are treated according to a "fast track" protocol, in most cases resulting in a hospital admission of only two days. This increases the chance that patient's release from hospital will be delayed due to wound drainage. The fact that our department recently started to perform hip and knee arthroplasty in a daycare setting increases this chance substantially.

In hemiarthroplasty of the knee, tissue adhesive was used in addition to conventional wound closure techniques with monocryl sutures. Resorbable monocryl sutures were used so that the usual visit to our outpatient department to remove the sutures was no longer necessary. However, we experienced an increase in wound drainage and complications using only monocryl. The addition of a tissue adhesive decreased the post-operative wound complication drastically. This in mind, we started to use tissue adhesive in regular hip and knee arthroplasty as well. With tissue adhesive in addition to conventional staples, we noticed good results. These results however, were subjective and not officially recorded.

In a previous study, good results are reported in decreasing wound drainage with the use of a tissue adhesive in addition to staples. Clinical relevance was not reported and the study design lacked a cost-effectiveness analysis (3) The increase in cost for the use of the tissue adhesive involved was noted by our board of directors. Because lack of a clear medical of financial benefit, we were asked to minimize the use of tissue adhesive, resulting in usage of tissue adhesive solely in a day care setting, which comprises only 5 to 10 percent of our treated population. Previous study reported a decrease in post-operative wound drainage when tissue adhesive was used in addition to staples in knee arthroplasty. However, no financial benefit is known, therefore this treatment has not been accepted into daily practice. In our department, prolonged hospital admission due to wound drainage is not found to be uncommon. Our hypothesis is that the addition of tissue adhesive in wound closure after hip and knee arthroplasty will significantly decrease post-operative wound drainage, leading to a reduced number of admission days. In addition, we expect less patients to return to our outpatient clinic for non-regular visits due to wound complications. Expensive bandages are used in our standard treatment protocol. Less wound drainage would mean less bandages. All these things combined will lead to a reduction in overall health care costs

ELIGIBILITY:
Inclusion Criteria:

* primary total hip or knee arthroplasty

Exclusion Criteria:

* revision surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: THA and TKA patients
Sampling Method: Probability Sample
Enrollment: 980 (Estimated)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-01-23 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Admission days | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Rutger van Geenen, MD, PhD, Principal Investigator — Amphia Hospital, Breda, the Netherlands
Locations (1):
- Amphia Hospital, Breda, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No